CLINICAL TRIAL: NCT00995709
Title: A 24 Week Multicenter, Randomized, Double-masked, Placebo Controlled Study to Assess the Difference in the Rate of Recurrent Exacerbations in Behçet¿s Patients With Posterior or Panuveitis Treated With AIN457 vs Placebo Adjunctive to Standard-of-care Immunosuppressive Therapy
Brief Title: Phase III Study in Refractory Behcet's Disease
Acronym: SHIELD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457C2303; 2009-011237-27 (EudraCT Number)
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Behcet Disease
Keywords: Behçet's disease,; intermediate uveitis; panuveitis; posterior uveitis; uveitis
MeSH Terms: conditions — Behcet Syndrome; Uveitis, Intermediate; Panuveitis; Uveitis, Posterior; Uveitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- AIN457C 300 mg every 2 week dosage regimen (Experimental): AIN457 300 mg was administered in 2 subcutaneous (s.c.) injections of 150 mg each. every 2 weeks
  Interventions: Drug: AIN457
- AIN457C 300 mg monthly dosage regimen (Experimental): AIN457 300 mg was administered in 2 subcutaneous (s.c.) injections of 150 mg e
  Interventions: Drug: AIN457
- Placebo (Placebo Comparator): Placebo was administered in 2 s.c. injections every 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457
  Arms: AIN457C 300 mg every 2 week dosage regimen
Drug: AIN457
  Arms: AIN457C 300 mg monthly dosage regimen
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this pivotal trial is to evaluate subcutaneous (SQ) AIN457 as an adjunctive therapy to reduce the rate of exacerbations of posterior uveitis or panuveitis secondary to Behçet's disease during the 24 weeks of study therapy as compared to standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Behçet's disease and with a history of recurrent uveitis in a least one eye.
* Documented evidence of >2 recurrent exacerbations of either intermediate uveitis, posterior uveitis or panuveitis in the study eye within the past 6 months (this could include the current exacerbation for patients having an acute exacerbation at screening). Exacerbations fulfilling the study inclusion criteria must have one or more of the following recorded in the patients patients medical record for each recurrent exacerbation:

  * >2+ vitreous haze with <2+ anterior chamber cell grade (intermediate or posterior uveitis) or >2+ vitreous haze with >2+ anterior chamber cell grade (panuveitis)
  * presence of retinal infiltrates or vasculitis or hemorrhages
  * documented >10 ETDRS letter or 2 line Snellen decrease in visual acuity attributed to ocular inflammation secondary to the recurrent exacerbation of Behçet's disease.
* Requirement for either of the following immunosuppressive therapies for at least 3 of the past 6 months for the treatment of or to prevent an exacerbation of ocular inflammation related to Behçet's disease:

  * Prednisone or equivalent >10 mg daily
  * The need for at least >1 periocular injection or >1 intravitreal corticosteroid injection in the study eye within the past 6 months (the last injection must have not been given within 6 weeks of screening)
  * Treatment with cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, mycophenolic acid or methotrexate either as monotherapy or in combination with or without steroids. (Patients treated at any time with chlorambucil or cyclophosphamide are not eligible for the study.)
* Patients not meeting the above specified criteria for immunomodulatory therapies are eligible for enrollment if they are intolerant to systemic immunomodulatory therapy as determined by the study investigator.

Exclusion Criteria:

* Subjects with infectious uveitis, uveitis due to other causes than Behçet's disease, or uveitis of unknown etiology.
* Less severe (i.e. anterior) uveitis associated with Behçet's disease.

Ocular treatments

* Treatment with intravitreal anti-VEGF agents administered to the study eye within 3 months prior to study screening.
* Treatment with any injected or implantable corticosteroid releasing device (i.e., flucinolone acetonide implant, Retisert®) in the study eye within the last 3 years.
* Intraocular surgery or laser photocoagulation in the study eye within the last 6 weeks prior to screening except for a diagnostic vitreous or aqueous tap with a small-gauge needle.

Systemic conditions or treatments

* Treatment with any live or live-attenuated vaccine (including vaccine for varicella-zoster virus or measles) within 2 months prior to screening.
* Any systemic biologic therapy (e.g. interferon, infliximab, daclizumab, etanercept, or adalimumab) given intravenously or subcutaneously within 3 months prior to screening and no prior treatment with AIN457.
* Any prior treatment with systemic alkylating agents (cyclophosphamide, chlorambucil).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (3):
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Houston, Texas
- Novartis Investigative Site, Alexandria, Egypt
- Novartis Investigative Site, Grenoble, France
- Germany (4):
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Münster
- Greece (8):
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Larissa, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Heraklion - Crete, GR
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- India (4):
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Angamaly
  - Novartis Investigative Site, New Delhi
- Israel (4):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (2):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
- Jordan (2):
  - Novartis Investigative Site, Amman
  - Novartis Investigative Site, Irbid
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (3):
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
- Switzerland (2):
  - Novartis Investigative Site, Lausanne, Switzerland
  - Novartis Investigative Site, Bern
- Novartis Investigative Site, Lin-Ko, Taiwan
- Tunisia (3):
  - Novartis Investigative Site, Monastir
  - Novartis Investigative Site, Sfax
  - Novartis Investigative Site, Tunis
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Altindag / Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

REFERENCES:
- [Derived] Dick AD, Tugal-Tutkun I, Foster S, Zierhut M, Melissa Liew SH, Bezlyak V, Androudi S. Secukinumab in the treatment of noninfectious uveitis: results of three randomized, controlled clinical trials. Ophthalmology. 2013 Apr;120(4):777-87. doi: 10.1016/j.ophtha.2012.09.040. Epub 2013 Jan 3. PMID 23290985

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457C 300 mg Every 2 Week Dosage Regimen: AIN457 300 mg was administered in 2 subcutaneous (s.c.) injections of 150 mg each.
- AIN457C 300 mg Monthly Dosage Regimen: AIN457 300 mg was administered in 2 subcutaneous (s.c.) injections of 150 mg each.
  One patient in the AIN457 300 mg monthly group (PID 0161/00002) was randomized; however, this patient did not meet eligibility criteria and never received study medication
- Placebo to AIN457C: Placebo was administered in 2 s.c. injections
Period: Overall Study
Arm/Group | AIN457C 300 mg Every 2 Week Dosage Regimen | AIN457C 300 mg Monthly Dosage Regimen | Placebo to AIN457C
Started | 39 | 40 | 39
Completed | 32 | 31 (patient in the 300 mg monthly group was randomized,was not eligible,never received study medication) | 34
Not Completed | 7 | 9 | 5
Not completed — Adverse Event | 4 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 4 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: a. One patient who screen-failed was inadvertently randomized to the AIN457 300 mg monthly group. This patient did not receive any study medication.
Groups:
- AIN457C 300 mg Monthly Dosage Regimen (a): AIN457 300 mg was administered in 2 subcutaneous (s.c.) injections of 150 mg each
- Total: Total of all reporting groups
Arm/Group | AIN457C 300 mg Every 2 Week Dosage Regimen | AIN457C 300 mg Monthly Dosage Regimen (a) | Placebo to AIN457C | Total
Number analyzed (Participants) | 39 | 40 | 39 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.2 (10.96) | 34.0 (11.86) | 32.5 (10.34) | 34.2 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 15 | 38
  Male | 27 | 29 | 24 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 39 | 39 | 37 | 115
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: Participants]
  France | 1 | 0 | 0 | 1
  Turkey | 19 | 18 | 18 | 55
  Germany | 1 | 1 | 1 | 3
  Greece | 3 | 5 | 4 | 12
  Italy | 3 | 2 | 2 | 7
  Spain | 1 | 0 | 1 | 2
  United States | 0 | 2 | 0 | 2
  Egypt | 1 | 2 | 2 | 5
  Israel | 2 | 0 | 1 | 3
  Jordan | 0 | 2 | 1 | 3
  Tunisia | 2 | 1 | 2 | 5
  Hong Kong | 1 | 1 | 1 | 3
  India | 1 | 2 | 1 | 4
  Korea, Republic Of | 2 | 4 | 4 | 10
  Singapore | 1 | 0 | 1 | 2
  Taiwan, Province Of China | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Recurrent Ocular Exacerbations in the Study Eye During 24 Weeks by Treatment
Time Frame: Baseline to week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Ocular Exacerbations
Arm/Group | AIN457C 300 mg Every 2 Week Dosage Regimen | AIN457C 300 mg Monthly Dosage Regimen (a) | Placebo to AIN457C
Number analyzed (Participants) | 39 | 39 | 39
Ocular Exacerbations | 7.7 (22.40) | 11.5 (28.19) | 7.7 (22.35)

2. Secondary Outcome: Change From Baseline for Composite Immunosuppressive Medication Score at Week 24 by Treatment (Full Analysis Set)
Description: For each corticosteroid medication, dose of the corticosteroid was first converted to a prednisone-equivalent dose. To determine the prednisone equivalent dose, the corticosteroid dose was multiplied by a conversion factor. . The total prednisone equivalent dose was calculated as the sum of the prednisone equivalent doses of all corticosteroids. Consequently, the total converted prednisone equivalent dose was used to obtain the immunosuppressive score. The key secondary efficacy variable was the change in total post-baseline immunosuppressive medication score from baseline.The score is actually the prednisoone equivalents taken by patient as calculated by conversion table. A reduction in prenisone or prenisone equivalents is a positive outcome. An increase in the number of prednisone equivalents suggests that the treatment is not efficacious or that there is disease progression. A score of 0 would be the lowest ( no steriods taken) and the upper limit is indeterminate.
Time Frame: 24 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: immunosuppressive medication score
Arm/Group | AIN457C 300 mg Every 2 Week Dosage Regimen | AIN457C 300 mg Monthly Dosage Regimen (a) | Placebo to AIN457C
Number analyzed (Participants) | 39 | 39 | 39
immunosuppressive medication score
  Baseline Score (n=39,39,39) | 7.769 (4.306) | 10.11 (5.3236) | 9.231 (3.8064)
  Week 24 (n=34,32,34) | 7.441 (4.4641) | 10.09 (5.3331) | 8.722 (3.2027)
  LOCF (n=39,39,39) | 7.769 (4.3036) | 10.11 (5.3236) | 9.231 (3.8064)

3. Secondary Outcome: To Determine the Effect of AIN457 on Macular Edema and Visual Acuity in Patients With Posterior Segment Uveitis Secondary to Behçet's Disease as Determined by Optical Coherence Tomography.
Description: Optical coherence tomography (OCT) is amedical imaging technique that uses light to capture micrometer-resolution, three-dimensional images from within optical scattering media (e.g., biological tissue). OCT is based on low-coherence interferometry, typically employing near-infrared light. The use of relatively long wavelength light allows it to penetrate into the scattering medium. OCT is a noninvasive procedure that uses optical interferometry to visualize the structures within the retina. Following dilation of the pupil, a light source operating at 850nm provides probe illumination which is split and detected with and without the refraction of the retinal tissues. Cross-sectional imaging is accomplished in 1.3 second by acquiring a sequence of interferometric A-scans. A false color tomogram of optical reflectivity is produced by the computer. Central foveal thickness will be the primary variable derived from OCT. A increase in thickness could translate to disease progression.
Time Frame: baseline, and wk 24 (end of study)
Population: (Full Analysis Set)
Measure: Mean (Standard Deviation); unit: change from baseline : micrometers
Arm/Group | AIN457C 300 mg Every 2 Week Dosage Regimen | AIN457C 300 mg Monthly Dosage Regimen (a) | Placebo to AIN457C
Number analyzed (Participants) | 39 | 39 | 39
change from baseline : micrometers | -26.5 (131.32) | 3.6 (75.29) | -49.4 (174.25)

4. Secondary Outcome: To Establish the Impact of AIN457 on Quality of Life of Posterior Segment Uveitis Patients Secondary to Behçet's Disease Refractory to Systemic Immunomodulatory Therapy as Measured by National Eye Institute Visual Function Questionaire-25 and Euroqol.
Description: The VFQ-25 is a reliable and valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ). It is especially useful in settings such as clinical trials, where interview length is a critical consideration. Scores range from 0 to 100, with higher scores indicating better visual function.
Time Frame: screening, and wk 24 (end of study)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AIN457C 300 mg Every 2 Week Dosage Regimen | AIN457C 300 mg Monthly Dosage Regimen (a) | Placebo to AIN457C
Number analyzed (Participants) | 39 | 39 | 39
Score
  Baseline (n= 38,35,39) | 62.46 (21.817) | 64.17 (25.549) | 62.11 (24.416)
  Week 24 (n=38,35,38) | 66.09 (24.295) | 73.68 (22.634) | 69.29 (21.858)

5. Secondary Outcome: To Observe the Effect of AIN457 on the Systemic Non-ocular Manifestations of Behçet's Disease in Patients With Posterior Segment Uveitis Requiring Systemic Immunosuppression as Measured by the Bechet's Disease Current Activity Form.
Description: The BDCAF scores oral and genital ulceration, skin, joint and gastrointestinal involvement, presence of fatigue and headache according to the duration of symptoms. The presence and type of large-vessel and central nervous system (CNS) involvement are documented. Eye activity was deemed present if there was a history of blurring of vision or if the eye was painful or red. . The BDCAF score was calculated by adding the score of each index and ranged between 0 and 12 A reduction in score signifies a lessening of the disease.
Time Frame: baseline and wk 24 (end of study)
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: change from baseline score
Arm/Group | AIN457C 300 mg Every 2 Week Dosage Regimen | AIN457C 300 mg Monthly Dosage Regimen (a) | Placebo to AIN457C
Number analyzed (Participants) | 16 | 17 | 19
change from baseline score | -1.3 (1.81) | -1.7 (1.49) | -1.1 (1.22)

6. Primary Outcome: Rate of Recurrent Ocular Exacerbations in the Study Eye During 24 Weeks by Treatment
Description: Patients number of occurences during a 24 week period.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | AIN457C 300 mg Every 2 Week Dosage Regimen | AIN457C 300 mg Monthly Dosage Regimen (a) | Placebo to AIN457C
Number analyzed (Participants) | 39 | 39 | 39
Participants
  0 recurrences | 15 | 15 | 11
  1 recurrence | 8 | 14 | 13
  2 recurrences | 8 | 3 | 5
  3 or more recurrences | 8 | 7 | 10

ADVERSE EVENTS:
Groups:
- AIN457 300mg Every 2 Weeks; AIN457 300mg Monthly: AIN457 300 mg was administered in 2 subcutaneous (s.c.) injections of 150 mg each.
- Placebo: Placebo was administered in 2 s.c. injections
Arm/Group | AIN457 300mg Every 2 Weeks | AIN457 300mg Monthly | Placebo
Serious Adverse Events (participants affected / at risk) | 6/39 | 8/39 | 5/39
Other Adverse Events (participants affected / at risk) | 28/39 | 25/39 | 22/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg Every 2 Weeks (N=39) | AIN457 300mg Monthly (N=39) | Placebo (N=39)
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Cataract cortical (Fellow eye) (Eye disorders) | 0 | 0 | 1
Cataract nuclear (Fellow eye) (Eye disorders) | 0 | 0 | 1
Cataract subcapsular (Fellow eye) (Eye disorders) | 0 | 0 | 1
Choroiditis (Fellow eye) (Eye disorders) | 1 | 0 | 0
Glaucoma (Fellow eye) (Eye disorders) | 0 | 0 | 1
Retinal infiltrates (Fellow eye) (Eye disorders) | 1 | 0 | 0
Retinal infiltrates (Study eye) (Eye disorders) | 1 | 0 | 0
Uveitis (Fellow eye) (Eye disorders) | 1 | 1 | 0
Uveitis (Study eye) (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Behcet's syndrome (Immune system disorders) | 0 | 1 | 0
Behcet's syndrome (Fellow eye) (Immune system disorders) | 0 | 1 | 0
Behcet's syndrome (Study eye) (Immune system disorders) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0
Hypopyon (Fellow eye) (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Intraocular pressure increased (Fellow eye) (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg Every 2 Weeks (N=39) | AIN457 300mg Monthly (N=39) | Placebo (N=39)
Cataract subcapsular (Fellow eye) (Eye disorders) | 3 | 1 | 0
Cataract subcapsular (Study eye) (Eye disorders) | 4 | 1 | 0
Eye pain (Study eye) (Eye disorders) | 1 | 2 | 2
Retinal vasculitis (Study eye) (Eye disorders) | 2 | 0 | 0
Vision blurred (Fellow eye) (Eye disorders) | 0 | 6 | 1
Vision blurred (Study eye) (Eye disorders) | 0 | 1 | 3
Visual acuity reduced (Study eye) (Eye disorders) | 4 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 2
Toothache (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 3
Fatigue (General disorders) | 2 | 2 | 4
Non-cardiac chest pain (General disorders) | 2 | 0 | 1
Oedema peripheral (General disorders) | 3 | 1 | 0
Pyrexia (General disorders) | 6 | 2 | 4
Conjunctivitis infective (Study eye) (Infections and infestations) | 1 | 2 | 1
Influenza (Infections and infestations) | 2 | 4 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Rash pustular (Infections and infestations) | 2 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Blood glucose increased (Investigations) | 0 | 2 | 0
Intraocular pressure increased (Study eye) (Investigations) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 9 | 6 | 9
Anxiety (Psychiatric disorders) | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial